CLINICAL TRIAL: NCT07153874
Title: The Effectiveness of a Physical Exercise Program in the Person Undergoing Cardiac Surgery
Brief Title: The Research Aims to Study the Effectiveness of a Physical Exercise Program on Indicators of Quality of Life and Functionality: It Will be Applied at Home to People Undergoing Cardiac Surgery, in Phase II of Cardiac Rehabilitation
Acronym: HeartBack2Beat
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Católica Portuguesa (Other)
Responsible Party: Principal Investigator, Pedro José Moreira Barbosa, PhD student, Universidade Católica Portuguesa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 115/2023
Record Dates: First submitted 2025-08-18; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Cardiac Surgery; Rehabilitation Program; Quality of Life; Functional Status

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental (Experimental): Group that will complete the structured and monitored physical exercise program.
  Interventions: Other: Physical exercise rehabilitation intervention
- Control (No Intervention): Group that receives no intervention during the study.

INTERVENTIONS:
Other: Physical exercise rehabilitation intervention — 12 weeks of physical exercise intervention, including aerobic snd anaerobic exercise at home. 36 sessions of monitorized training with distance supervision.
  Other Names: HeartBackToBeat
  Arms: Experimental

SUMMARY:
The goal of this clinical trial is to test the effectiveness of an physical exercise intervention in people after cardiac surgery, namely valve replacement and coronary artery bypass graft. The main question[s] it aims to answer are: • what is the influence of a physical exercise program on quality of life in people after cardiac surgery • what is the influence of a physical exercise program on functional status in people after cardiac surgery. Participants will be allocated to exepriemtal group and perform a physical exercise program during 12 weeks and the program is composed by aerobic and anaerobic exercise. They will be evaluated at the beginning, middle and in the end of the program. Researchers will compare the experimental and the control group to see the effects in quality of life and functional status.

ELIGIBILITY:
* Clients undergoing cardiac surgery for the first time: heart valve surgery, coronary artery bypass grafting, after discharge from hospital in a home setting;
* Clients at low and moderate risk of cardiovascular events;
* Clients over the age of 18;
* Clients who are part of the localities assisted by the hospital unit;
* Clients with preserved cognitive capacity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2024-02-19 (Actual); Primary Completion 2024-06-10 (Actual); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Functionality | The results are expected to be measured at the beginning of the program, at six weeks, and at the end (at 12 weeks).
  Functionality is the ability regarding basic physical and cognitive activities such as walking or reaching, focusing attention, and communicating, as well as the routine activities of daily living, including eating, bathing, dressing, transferring, and toileting; and life situations such as school or play for children and, for adults, work outside the home or maintaining a household. It will be measured by the London Chest Daily Activities scale.
Perceived Quality of life | The results are expected to be measured at the beginning of the program, at six weeks, and at the end (at 12 weeks).
  Quality of life is a generic concept reflecting concern with the modification and enhancement of life attributes, e.g., physical, political, moral, social environment as well as health and disease. It will be measured by the Short Form-36 quality of life assessment scale.
Tolerance to physical exercise | The results are expected to be measured at the beginning of the program, at six weeks, and at the end (at 12 weeks).
  Tolerance to physical exercise is the exercise capacity of an individual as measured by endurance (maximal exercise duration and/or maximal attained work load) during an exercise test. It will be measured by the 6-minute walk test.

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Hospitalar Universitário de São João, Porto, Porto District, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] American College of Sports and Medicine. (2021). Guidelines for Exercise Testing and Prescription (W. Kluwer Ed. 11 ed.). Philadelphia
- [Background] Piepoli MF, Corra U, Benzer W, Bjarnason-Wehrens B, Dendale P, Gaita D, McGee H, Mendes M, Niebauer J, Zwisler AD, Schmid JP; Cardiac Rehabilitation Section of the European Association of Cardiovascular Prevention and Rehabilitation. Secondary prevention through cardiac rehabilitation: from knowledge to implementation. A position paper from the Cardiac Rehabilitation Section of the European Association of Cardiovascular Prevention and Rehabilitation. Eur J Cardiovasc Prev Rehabil. 2010 Feb;17(1):1-17. doi: 10.1097/HJR.0b013e3283313592. PMID 19952757
- [Background] Rossello X, Dorresteijn JA, Janssen A, Lambrinou E, Scherrenberg M, Bonnefoy-Cudraz E, Cobain M, Piepoli MF, Visseren FL, Dendale P, This Paper Is A Co-Publication Between European Journal Of Preventive Cardiology European Heart Journal Acute Cardiovascular Care And European Journal Of Cardiovascular Nursing. Risk prediction tools in cardiovascular disease prevention: A report from the ESC Prevention of CVD Programme led by the European Association of Preventive Cardiology (EAPC) in collaboration with the Acute Cardiovascular Care Association (ACCA) and the Association of Cardiovascular Nursing and Allied Professions (ACNAP). Eur J Prev Cardiol. 2019 Sep;26(14):1534-1544. doi: 10.1177/2047487319846715. Epub 2019 Jun 24. PMID 31234648
- [Background] Supervia M, Medina-Inojosa J, Martinez-Jarreta B, Lopez-Jimenez F, Vickers K, Terzic CM, Thomas RJ. Cardiac Rehabilitation Completion Study: Barriers and Potential Solutions. J Cardiopulm Rehabil Prev. 2022 Sep 1;42(5):375-377. doi: 10.1097/HCR.0000000000000709. No abstract available. PMID 36044761
- [Background] Thomas RJ, King M, Lui K, Oldridge N, Pina IL, Spertus J; American Association of Cardiovascular and Pulmonary Rehabilitation/American College of Cardiology/American Heart Association Cardiac Rehabilitation/Secondary Prevention Performance Measures Writing Committee. AACVPR/ACC/AHA 2007 performance measures on cardiac rehabilitation for referral to and delivery of cardiac rehabilitation/secondary prevention services. Circulation. 2007 Oct 2;116(14):1611-42. doi: 10.1161/CIRCULATIONAHA.107.185734. Epub 2007 Sep 20. No abstract available. PMID 17885210
- [Background] Thomas RJ, Balady G, Banka G, Beckie TM, Chiu J, Gokak S, Ho PM, Keteyian SJ, King M, Lui K, Pack Q, Sanderson BK, Wang TY. 2018 ACC/AHA Clinical Performance and Quality Measures for Cardiac Rehabilitation: A Report of the American College of Cardiology/American Heart Association Task Force on Performance Measures. J Am Coll Cardiol. 2018 Apr 24;71(16):1814-1837. doi: 10.1016/j.jacc.2018.01.004. Epub 2018 Mar 29. No abstract available. PMID 29606402
- [Background] Vidal-Almela S, Czajkowski B, Prince SA, Chirico D, Way KL, Pipe AL, Reed JL. Lessons learned from community- and home-based physical activity programs: A narrative review of factors influencing women's participation in cardiac rehabilitation. Eur J Prev Cardiol. 2021 Jul 10;28(7):761-778. doi: 10.1177/2047487320907748. PMID 33611528